CLINICAL TRIAL: NCT05059275
Title: Study on Pathogenesis and Treatment of Sacral Tarlov Cysts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Yuntao Lu, Professor, Southern Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMU-Neurosurgery-spine
Record Dates: First submitted 2021-09-11; First posted 2021-09-28 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Tarlov Cysts
Keywords: Sacral perineural cyst; Tarlov cyst; Ostium closure; Surgical treatment
MeSH Terms: conditions — Tarlov Cysts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified operation group (Experimental): Undergo the modified ostium obstruction surgery due to symptomatic TCs.
  Interventions: Procedure: modified ostium obstruction surgery

INTERVENTIONS:
Procedure: modified ostium obstruction surgery — An ostium at the end of the site where the nerve root enters the dural sac, from which CSF could flow continuously along the subarachnoid space, was identified An appropriate amount of autologous soft adipose tissue was removed under the skin of the incision or deep in the upper part of the buttock (Iliac spine incision, for less subcutaneous fat patients). It was then trimmed to resemble a gourd or dumbbell, with a relatively small middle section and two relatively large end sections. Trimmed graft was inserted into the neck of the sac and subarachnoid space below the dural sac so that it plugs the ostium inside and outside After filling the graft, Prolene 6-0 was used to continuously suture and close the ostium and dural sac starting from the lower part of the nerve root sheath and the ostium.The residual cyst cavity filled with autologous fat and gelatin sponge

SUMMARY:
The pathogenesis of sacral Tarlov cysts (TCs) is still unclear. In this study, histological techniques were used to clarify the anatomical membranous layers of TCs and further explore the pathogenesis of them.Although many approaches have been used to treat TCs, there is no consensus on the optimal treatment. Microsurgery is now increasingly recommended as the preferred treatment with the best long-term outcomes.However, some authors have proposed the opposite view because current microsurgical techniques fail to completely close the ostium between the cyst and subarachnoid space.Consequently, could lead to leakage of cerebrospinal fluid, pseudomeningocele , or a high frequency of cysts recurrence, which are the main reasons for surgical failure and also the biggest scruple when microsurgery is chosen. Herein, we present a new method of cyst separation and ostium closure, and evaluate its clinical reliability and effectiveness for surgical treatment of Tarlov cysts through the prospective study.

DETAILED DESCRIPTION:
1. Part of the intact cyst wall was removed under the microscope and fixed in 10% formalin solution. After dehydration and paraffin embedding, tissue sections (thickness: 6μm) were prepared and dewaxed to water. Sirius red stain drops were stained for 1 hour. The staining liquid on the surface of the slices was removed after a little flushing with water. The slices were dehydrated and transparent, sealed with neutral gum, and the membranous layers of the capsule walls were observed under a microscope.It has been observed in previous surgeries that all cysts were incompressible and remained filled after opening the distal wall of the cyst to release cerebrospinal fluid（CSF). These findings lent support for the proposed valve mechanism as the etiology of the entity becoming symptomatic. In this study, the cyst was observed in the following way: the dural sac was opened to expose the ostium to observe whether the cystic fluid would reverse outflow and shrink the cyst; In this way, the existence of a "one-way valve" can be further verified.
2. Modified microsurgical method is used to treat patients who met the inclusion criteria. To evaluate the surgical effect, we record and statistically compare the patients'outcomes before surgery and at the postoperative follow-up, which include the following: 1) Demographic data: sex, age, height, weight, body mass index (BMI), etc.; 2) clinical manifestations: symptoms and their features, complications, and long-term recovery; 3) Imaging findings: maximum diameter, location, shape, number, intracapsular nerve root condition, and postoperative outcome of TCs. 4) Surgical characteristics: operative process and time, intraoperative blood loss, assistive technologies, etc.; 5) Neurologic assessment using the following tools: The visual analogue scale (VAS), Scoring System for the Clinical Evaluation of Patients with Spinal Processes (hereinafter referred to as SCPS), Oswestry Disability Index (ODI), Japanese Orthopedic Association Scores 29 (JOA), and modified evaluation criteria for the efficacy of lumbar function (MacNab).All patients are required to return for MRI review and neurofunctional assessment at 3 and 12 months postoperatively, followed by annual examinations thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Conform to the surgical indications and undergo modified microscopic surgery in our department;
* Undergo regular review and long-term clinical effect evaluation;
* Agree to participate in this study.

Exclusion Criteria:

* Ineligible for modified microscopic surgery or unwilling to undergo it;
* Failure to cooperate with follow-up work or lost to follow-up；
* Did not agree to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2022-09-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
The visual analogue scale (VAS) | Three months after surgery
  The visual analogue scale (VAS)，Score range: 0-10, with a higher score indicating more severe pain
Scoring System for the Clinical Evaluation of Patients with Spinal Processes | One year after surgery
  Scoring System for the Clinical Evaluation of Patients with Spinal Processes (hereinafter referred to as SCPS)，score range：0- 25.The higher the score, the better the spinal cord function state.
Evaluation of imaging results (magnetic resonance and computerized tomography) | One days before surgery
  Maximum diameter of TCs.
Histological examination results | One day after surgery
  Part of the intact cyst wall was stained with Sirius red and its anatomical membranous layers were observed under a microscope.

SECONDARY OUTCOMES:
Surgical characteristics | During surgery
  Operating time
Clinical manifestations | Two days before surgery
  Duration of symptoms
Demographic data | Three days before surgery
  Age

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From the completion of data collection to 1 month after the publication of the article

REFERENCES:
- [Background] Sharma M, SirDeshpande P, Ugiliweneza B, Dietz N, Boakye M. A systematic comparative outcome analysis of surgical versus percutaneous techniques in the management of symptomatic sacral perineural (Tarlov) cysts: a meta-analysis. J Neurosurg Spine. 2019 Feb 8;30(5):623-634. doi: 10.3171/2018.10.SPINE18952. Print 2019 May 1. PMID 30738394
- [Background] Singh PK, Singh VK, Azam A, Gupta S. Tarlov cyst and infertility. J Spinal Cord Med. 2009;32(2):191-7. doi: 10.1080/10790268.2009.11760771. PMID 19569467
- [Background] Fletcher-Sandersjoo A, Mirza S, Burstrom G, Pedersen K, Kuntze Soderqvist A, Grane P, Fagerlund M, Edstrom E, Elmi-Terander A. Management of perineural (Tarlov) cysts: a population-based cohort study and algorithm for the selection of surgical candidates. Acta Neurochir (Wien). 2019 Sep;161(9):1909-1915. doi: 10.1007/s00701-019-04000-5. Epub 2019 Jul 3. PMID 31270612
- [Background] Liu B, Wang Z, Lin G, Zhang J. Radiculoplasty with reconstruction using 3D-printed artificial dura mater for the treatment of symptomatic sacral canal cysts: Two case reports. Medicine (Baltimore). 2018 Dec;97(49):e13289. doi: 10.1097/MD.0000000000013289. PMID 30544388
- [Background] Guo D, Shu K, Chen R, Ke C, Zhu Y, Lei T. Microsurgical treatment of symptomatic sacral perineurial cysts. Neurosurgery. 2007 Jun;60(6):1059-65; discussion 1065-6. doi: 10.1227/01.NEU.0000255457.12978.78. PMID 17538380
- [Background] ABBOTT KH, LEIMBACH WH, RETTER RH. The role of perineurial sacral cysts in the sciatic and sacrococcygeal syndromes; a review of the literature and report of 9 cases. J Neurosurg. 1957 Jan;14(1):5-21. doi: 10.3171/jns.1957.14.1.0005. No abstract available. PMID 13385699